CLINICAL TRIAL: NCT00657202
Title: Pilot Study of Ranibizumab (Lucentis) for Neurofibromas Associated With Neurofibromatosis 1
Brief Title: Ranibizumab for Neurofibromas Associated With Neurofibromatosis 1
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Scott Randall Plotkin, MD, PhD, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-332
Record Dates: First submitted 2008-03-27; First posted 2008-04-14 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Neurofibromatosis Type 1; Cutaneous Neurofibromas
Keywords: NF1; neurofibroma; ranibizumab; Lucentis
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Given as an injection into three cutaneous neurofibromas on day 1 of the study treatment.
  Other Names: Lucentis

SUMMARY:
The purpose of this research study is to determine if ranibizumab can prevent the growth of neurofibromas. We will also be collecting extra blood and serum samples to help us learn more about NF1. Ranibizumab is a drug that affects the development of blood vessels that feed tumors. It targets a substance in the body called VEGF (Vascular Endothelial Growth Factor). VEGF helps tumors to grow and survive by supporting the growth of blood vessels that bring nutrients to the tumor. VEGF is made by cancerous tumors and also by non-cancerous tumors such as neurofibromas.

DETAILED DESCRIPTION:
* Participants will receive one injection of ranibizumab into 3 tumors on their skin (one dose per tumor) on day 1 of treatment. One other tumor will be injected with normal saline solution. The saline solution-called a control-is necessary to determine whether injections (without medicine) can cause a tumor to shrink. Tumors will be measured and photographed prior to treatment. Ranibizumab tumors will be removed on days 8, 15, and 29; the saline treated tumor will be removed on day 29.
* Participants will come into the clinic once a week for a total of 4 weeks and then again on Days 35. 57 and 85 for post-treatment visits. Some of the following tests and procedures will be performed: physical examination (including photographs of tumors), review of current medications, vital signs, routine blood tests, serum chemistry blood tests, interstitial fluid pressure measurements and tumor samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have diagnosis of NF1 based on NIH criteria with two or more of the following characteristics: a) Six or more cafe-au-lait macules b) Skin fold freckling in the axilla or groin c) Optic pathway glioma d) Two or more Lisch nodules of the iris e) Distinctive bony lesions such as dysplasia of the sphenoid wing or of a long bone such as the tibia f) Two or more neurofibromas of any type or 1 or more plexiform neurofibroma g) First degree relative with NF1
* At least four cutaneous neurofibromas on skin exam with the following qualities: a) the lesion must be discrete by clinical exam and must be at least 5mm away from another skin tumor b) the lesion must be amenable to measurement with calipers with minimum dimension of 5mm and maximum dimension of 20mm c)the lesions cannot be located on the face, scalp, or groin and must be located in an area that can be photographed d) histologic confirmation of tumor type is not required in the setting of compatible clinical setting
* Must be willing to have treated CNF surgically removed during the study
* 18 years of age or older
* Normal organ and marrow function as described in the protocol

Exclusion Criteria:

* Pregnant or breast-feeding women
* Chemotherapy or radiotherapy within 6 weeks prior to entering the study
* Receiving any other investigational agent
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as ranibizumab
* Hypertension that cannot be controlled by medications
* Known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhages in the past
* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting the study treatment
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Determine the effect of inhibiting VEGF signaling on tumor volume and tumor interstitial fluid pressure by local injection of ranibizumab into cutaneous neurofibromas. | 2 years

SECONDARY OUTCOMES:
To identify angiogenic molecules upregulated in neurofibromas treated with ranibizumab. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Plotkin, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States